CLINICAL TRIAL: NCT02023697
Title: A Three Arm Randomized, Open-label Phase II Study of Radium-223 Dichloride 50 kBq/kg (55 kBq/kg After Implementation of NIST Update) Versus 80 kBq/kg (88 kBq/kg After Implementation of NIST Update), and Versus 50 kBq/kg (55 kBq/kg After Implementation of NIST Update) in an Extended Dosing Schedule in Subjects With Castration-resistant Prostate Cancer Metastatic to the Bone
Brief Title: Standard Dose Versus High Dose and Versus Extended Standard Dose Radium-223 Dichloride in Castration-resistant Prostate Cancer Metastatic to the Bone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16507; 2013-003118-42 (EudraCT Number)
Record Dates: First submitted 2013-12-24; First posted 2013-12-30 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-06

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Radium-223 dichloride (Standard dose) (Experimental): One injection to be administered every 4 weeks up to 6 injections. The dose per injection is 50 kBq/kg body weight (55 kBq/kg after implementation of NIST update).
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
- Radium-223 dichloride (High dose) (Experimental): One injection to be administered every 4 weeks up to 6 injections. The dose per injection is 80 kBq/kg body weight (88 kBq/kg after implementation of NIST update).
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
- Radium-223 dichloride (Extended standard dose) (Experimental): One injection to be administered every 4 weeks up to 12 injections. The dose per injection is 50 kBq/kg body weight (55 kBq/kg after implementation of NIST update).
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

SUMMARY:
This study will assess different doses and regimens of radium-223 dichloride on the incidence of symptomatic skeletal events. Eligible subjects must have castration resistant prostate cancer with 2 or more skeletal metastases documented within 8 weeks of randomization. Subjects will be randomized to one of 3 treatment arms in a 1:1:1 fashion: a standard regimen of radium-223 dichloride of 50 kBq/kg (55 kBq/kg after implementation of NIST update) injections every month for 6 months, a high dose regimen of 80 kBq/kg (88 kBq/kg after implementation of NIST update)injections every month for 6 months or an extended duration regimen of 50 kBq/kg (55 kBq/kg after implementation of NIST update) injections every month for 12 months. Following the treatment phase, subjects will be followed up every 12 weeks for a minimum of 2 years, at which point they will enter a long term follow-up period during which they are seen every 6 months for up to 7 years after the last dose of radium dichloride. Symptomatic skeletal event and safety endpoints will be assessed at each clinic visit. Pain and analgesic use data will be collected every 4 weeks through Week 48. Additionally, radiological assessments including MRI/CT of the abdomen and pelvis and chest CT, as well as technetium-99 bone scans will be performed at Weeks 8, 16, and 24 and continue every 12 weeks thereafter until disease progression is documented in either the bone or in soft tissue. Radiological imaging will be evaluated by blinded central review.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Castration-resistant disease defined as:

  * Serum testosterone level: ≤ 50 ng/dL (1.7 nmol/L)
  * Bilateral orchiectomy or maintenance on androgen ablation therapy with luteinizing-hormone-releasing hormone (LHRH) agonist or antagonist, or polyestradiol phosphate
  * Serum PSA (Prostate specific antigen) progression defined as 2 subsequent increases in PSA over a previous reference value (a minimum of 2 ng/mL [μg/L]) OR
  * Radiographic evidence of disease progression in bone (according to Prostate Cancer Clinical Trials Working Group 2 [PCWG2] criteria) with or without PSA progression
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0 to 2. In case of ECOG PS 2, the PS has to be due to metastatic prostate cancer to the bone.
* Two or more skeletal metastases (≥ 2 hot spots) on bone scintigraphy within 8 weeks of randomization

Exclusion Criteria:

* History of visceral metastasis, or visceral metastases
* Lymphadenopathy with lymph nodes exceeding 3 cm in short axis diameter
* Central nervous system (CNS) metastases
* Treatment with cytotoxic chemotherapy for prostate cancer within the previous 4 weeks prior to randomization, or planned treatment with cytotoxic chemotherapy agents for prostate cancer during the treatment period or follow-up
* Chronic conditions associated with non-malignant abnormal bone growth (e.g. confirmed Paget's disease of bone)
* Prior treatment with radium-223 dichloride
* Prior systemic radiotherapy and hemibody external radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (65):
- United States (12):
  - Scottsdale, Arizona
  - New Haven, Connecticut
  - Fort Myers, Florida
  - Bethesda, Maryland
  - Rockville, Maryland
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - East Setauket, New York
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
- Australia (5):
  - Adelaide, South Australia
  - Melbourne, Victoria
  - Box Hill
  - Darlinghurst
  - Westmead
- Brazil (5):
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo
  - IBCC - Instituto Brasileiro de Controle do Cancer, São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
- Canada (4):
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Santiago, Chile
- Czechia (2):
  - Chomutov
  - Prague
- France (3):
  - Nantes
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (3):
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Dresden, Saxony
- Israel (6):
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
- Italy (4):
  - Meldola, Emilia-Romagna
  - Rome, Lazio
  - Turin, Piedmont
  - Arezzo, Tuscany
- South Korea (3):
  - Busan, Busan Gwang''yeogsi
  - Seoul, Seoul Teugbyeolsi
  - Seoul
- Spain (5):
  - L'Hospitalet de Llobregat, Barcelona
  - Palma de Mallorca, Illes Baleares
  - Barcelona
  - Madrid
  - Pamplona
- Sweden (4):
  - Gothenburg
  - Karlstad
  - Sundsvalls
  - Umeå
- Taiwan (5):
  - Taipei City, Taipei
  - Guishan Township, Taoyuan
  - Kaohsiung City
  - Taichung
  - Taipei
- United Kingdom (3):
  - Bebington, Merseyside
  - Taunton, Somerset
  - Northwood

REFERENCES:
- [Derived] Sternberg CN, Saad F, Graff JN, Peer A, Vaishampayan UN, Leung E, Rosenbaum E, Gurney H, Epstein RJ, Davis ID, Wu B, Trandafir L, Wagner VJ, Hussain M. A randomised phase II trial of three dosing regimens of radium-223 in patients with bone metastatic castration-resistant prostate cancer. Ann Oncol. 2020 Feb;31(2):257-265. doi: 10.1016/j.annonc.2019.10.025. Epub 2019 Dec 23. PMID 31959342

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 391 participants assigned to treatment in the intention to treatment (ITT) analysis set, 370 participants (94.6%) received at least one dose of radium-223 dichloride, and a total of 21 participants (5.4%) never received treatment
Groups:
- Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride (Xofigo, BAY88-8223) 55 kBq/kg intravenously (IV) every 28 days for up to 6 doses ("standard dose"). Participants who discontinued study treatment and who did not have an SSE entered an active follow-up period with clinic visits. Participants from the treatment period or the active follow-up period with clinic visits who could no longer travel entered an active follow-up period without clinic visits. All study participants eligible for further follow-up were either in this study or in a separate long term follow-up study for up to 7 years.
- Radium-223 Dichloride 88 kBq/kg, 6 Doses (Arm B): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride (Xofigo, BAY88-8223) 88 kBq/kg IV every 28 days for up to 6 doses ("high dose"). Participants who discontinued study treatment and who did not have an SSE entered an active follow-up period with clinic visits. Participants from the treatment period or the active follow-up period with clinic visits who could no longer travel entered an active follow-up period without clinic visits. All study participants eligible for further follow-up were either in this study or in a separate long term follow-up study for up to 7 years.
- Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride (Xofigo, BAY88-8223) 55 kBq/kg IV every 28 days for up to 12 doses ("extended dose"). Participants who discontinued study treatment and who did not have an SSE entered an active follow-up period with clinic visits. Participants from the treatment period or the active follow-up period with clinic visits who could no longer travel entered an active follow-up period without clinic visits. All study participants eligible for further follow-up were either in this study or in a separate long term follow-up study for up to 7 years.
Period: Treatment Period
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 88 kBq/kg, 6 Doses (Arm B) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Started (Randomized, Intent-To-Treatment (ITT)) | 130 | 130 | 131
Received Treatment | 125 | 124 | 121
Completed | 84 | 67 | 29
Not Completed | 46 | 63 | 102
Not completed — Radiological progression | 13 | 17 | 26
Not completed — Never Treated | 5 | 6 | 10
Not completed — Adverse Event | 13 | 25 | 23
Not completed — Logistical difficulties | 1 | 1 | 1
Not completed — Clinical progression | 10 | 8 | 28
Not completed — Withdrawal by Subject | 4 | 5 | 13
Not completed — Safety outcome reached | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Period: Active Follow-up Period
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 88 kBq/kg, 6 Doses (Arm B) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Started (Entered active follow-up) | 120 (Not all participants in ITT entered active follow-up.) | 120 (Not all participants in ITT entered active follow-up.) | 116 (Not all participants in ITT entered active follow-up.)
Completed | 28 | 21 | 17
Not Completed | 92 | 99 | 99
Not completed — Withdrawal by Subject | 5 | 13 | 7
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Deterioration of general condition | 1 | 1 | 1
Not completed — Other unspecified | 2 | 0 | 1
Not completed — Clinical progression | 0 | 2 | 1
Not completed — Radiological progression | 0 | 0 | 1
Not completed — Death | 83 | 82 | 87
Period: Long-term Follow-up Period
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 88 kBq/kg, 6 Doses (Arm B) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Started | 28 | 21 | 17
Completed | 0 | 0 | 0
Not Completed | 28 | 21 | 17
Not completed — Death | 9 | 6 | 4
Not completed — Withdrawal by Subject | 6 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Entered the long-term follow-up study | 6 | 9 | 6
Not completed — Technical problems | 0 | 0 | 1
Not completed — Other unspecified | 6 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 88 kBq/kg, 6 Doses (Arm B) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C) | Total
Number analyzed (Participants) | 130 | 130 | 131 | 391
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (8.6) | 70.9 (8.3) | 70.0 (8.1) | 70.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 130 | 130 | 131 | 391
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 6 | 10
  Not Hispanic or Latino | 125 | 124 | 120 | 369
  Unknown or Not Reported | 4 | 3 | 5 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 104 | 102 | 108 | 314
  Black or African American | 3 | 5 | 5 | 13
  Asian | 17 | 17 | 13 | 47
  Not reported | 6 | 6 | 5 | 17
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance status (ECOG PS): 0-Fully active, able to carry on all pre-diseases performance without restriction, (Karnofsky 90-100); 1- Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature,(Karnofsky 70-80) 2-Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours. (Karnofsky 50-60); 3-Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. (Karnofsky 30-40); 4-Completely disabled.
  Participants
    0 | 48 | 59 | 49 | 156
    1 | 78 | 67 | 77 | 222
    2 | 4 | 4 | 5 | 13
Average Worst Pain Score (WPS) [Mean (Standard Deviation); unit: scores on a scale] — Brief Pain Short Form (BPI-SF) encompasses 4 different items to capture the variability of pain over time (pain at its "worst," "least," "average," and "now"). For this study, only the worst pain score (WPS) in the last 24 hours was assessed (a visual analogic scale ranging 0-10, with 0 meaning "no pain" and 10 meaning "pain as bad as you can imagine"), and the mean score of the 7 days prior to the study visit or telephone contact was calculated and this value was recorded in the participant's reported outcome pain data. Population: The last assessment collected prior to randomization was used as baseline value. If no assessment was done prior to randomization, then the assessment collected after randomization but prior to first dose was used as baseline. Number of analyzed reflect the participants with data available at baseline.
  scores on a scale
    number analyzed (Participants) | 128 | 125 | 122 | 375
    (all) | 3.6 (2.6) | 3.3 (2.5) | 3.4 (2.6) | 3.4 (2.5)
Extent of disease [Count of Participants; unit: Participants]
  Normal or abnormal because of benign bone disease | 0 | 1 | 0 | 1
  <6 metastases | 19 | 22 | 19 | 60
  6-20 metastases | 52 | 53 | 52 | 157
  >20 lesions but not a superscan | 47 | 48 | 54 | 149
  Superscan | 12 | 6 | 6 | 24
Time from initial prostate cancer diagnosis to randomization [Median (Full Range); unit: months] | 58.9 [2 to 285] | 72.9 [7 to 279] | 67.1 [8 to 396] | 66.8 [2 to 396]
Time from initial bone metastases diagnosis to randomization [Median (Full Range); unit: months] | 30.8 [2 to 231] | 29.9 [1 to 170] | 37.5 [1 to 397] | 31.7 [1 to 397]
Time from most recent prostate cancer progression to randomization [Median (Full Range); unit: months] — Population: The last assessment collected prior to randomization was used as baseline value. If no assessment was done prior to randomization, then the assessment collected after randomization but prior to first dose was used as baseline. Number of analyzed reflect the participants with data available at baseline.
  months
    number analyzed (Participants) | 129 | 130 | 131 | 390
    (all) | 1.4 [0 to 8] | 1.4 [0 to 9] | 1.3 [0 to 10] | 1.3 [0 to 10]
Time from most recent bone metastases progression to randomization [Median (Full Range); unit: months] — Population: The last assessment collected prior to randomization was used as baseline value. If no assessment was done prior to randomization, then the assessment collected after randomization but prior to first dose was used as baseline. Number of analyzed reflect the participants with data available at baseline.
  months
    number analyzed (Participants) | 118 | 119 | 121 | 358
    (all) | 2.3 [0 to 34] | 2.8 [0 to 93] | 1.9 [0 to 41] | 2.4 [0 to 93]
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: The last assessment collected prior to randomization was used as baseline value. If no assessment was done prior to randomization, then the assessment collected after randomization but prior to first dose was used as baseline. Number of analyzed reflect the participants with data available at baseline.
  kg/m^2
    number analyzed (Participants) | 126 | 127 | 124 | 377
    (all) | 28.4 (5.2) | 28.0 (5.2) | 29.1 (5.4) | 28.5 (5.3)
Time from first bone metastases progression to most recent progression [Median (Full Range); unit: months] — Population: The last assessment collected prior to randomization was used as baseline value. If no assessment was done prior to randomization, then the assessment collected after randomization but prior to first dose was used as baseline. Number of analyzed reflect the participants with data available at baseline.
  months
    number analyzed (Participants) | 118 | 119 | 120 | 357
    (all) | 7.9 [0 to 72] | 8.9 [0 to 71] | 13.4 [0 to 120] | 9.5 [0 to 120]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Event Defining SSE Free Survival - High Dose vs. Standard Dose
Description: Symptomatic skeletal event (SSE) free survival is based on the following events: the use of external beam radiotherapy (EBRT) to relieve skeletal symptoms; the occurrence of new symptomatic pathological bone fractures (vertebral or nonvertebral); the occurrence of spinal cord compression; a tumor related orthopedic surgical intervention, and death. In this evaluation - comparison 1, SSE-FS following randomization is defined in ITT participants as the time from randomization to an SSE or death, whichever occurs first.
Time Frame: From randomization to 135 SSE-FS events have been observed in comparison 1 or 75 SSE-FS events observed in comparison 2, whichever occurred last (approximately 36 months from first patient randomization)
Population: Intent-to-treat (ITT): All randomized participants. Data from Arm C are truncated at 7th dose date when pooling with Arm A, therefore Pooled Arm A+C included 261 participants.
Measure: Count of Participants; unit: Participants
Groups:
- Radium-223 88 kBq/kg, 6 Doses (Arm B): Participants who were randomized in a 1:1:1 fashion received radium-223 dichloride 88 kBq/kg IV every 28 days for up to 6 doses ("high dose").
- Pooled Radium-223 55 kBq/kg (Arms A and C): Pooled Arms A and C, participants who were randomized in a 1:1:1 fashion received radium-223 dichloride 55 kBq/kg IV every 28 days for up to 6 and 12 doses, respectively.
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
Participants | 85 | 118

2. Primary Outcome: Symptomatic Skeletal Event-Free Survival - High Dose vs. Standard Dose
Description: In this evaluation - comparison 1, SSE-FS following randomization is defined in ITT participants as the time from randomization to an SSE or death, whichever occurs first.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
months | 12.9 [10.9 to 14.8] | 12.3 [10.3 to 13.5]
Statistical Analysis 1: Comparison: Radium-223 88 kBq/kg, 6 Doses (Arm B) vs Pooled Radium-223 55 kBq/kg (Arms A and C); Test type: Other; p = 0.7047, Log Rank; Hazard Ratio (HR) = 1.057, 80% CI 2-sided [0.878 to 1.272] — Arm B / Arm (A+C)

3. Primary Outcome: Number of Participants With an Event Defining SSE Free Survival - Extended Dose vs. Standard Dose
Description: Symptomatic skeletal event (SSE) free survival is based on the following events: the use of external beam radiotherapy (EBRT) to relieve skeletal symptoms; the occurrence of new symptomatic pathological bone fractures (vertebral or nonvertebral); the occurrence of spinal cord compression; a tumor related orthopedic surgical intervention, and death. In this evaluation - Comparison 2, SSE-FS from 6th dose is defined in W24 participants as the time from Week 24 baseline (the 6th dose date) to an SSE or death, whichever occurs first.
Time Frame: as for outcome 1
Population: Week 24 (W24): All ITT participants in Arm A (standard dose) and Arm C (extended dosing) treated with radium-223 dichloride and eligible for further treatment at W24 (i.e., 7th injection). All participants who received 6 doses from Arm A and participants who received >=6 doses from Arm C were included .
Measure: Count of Participants; unit: Participants
Groups:
- Radium-223 55 kBq/kg, 6 Doses (Arm A): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride 55 kBq/kg IV every 28 days for up to 6 doses ("standard dose").
- Radium-223 88 kBq/kg, 12 Doses (Arm C): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride 55 kBq/kg IV every 28 days for up to 12 doses ("extended dose").
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
Participants | 41 | 40

4. Primary Outcome: Symptomatic Skeletal Event-Free Survival - Extended Dose vs. Standard Dose
Description: In this evaluation - Comparison 2, SSE-FS from 6th dose is defined in W24 participants as the time from Week 24 baseline (the 6th dose date) to an SSE or death, whichever occurs first.
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Median (80% Confidence Interval); unit: months
Groups:
- Radium-223 88 kBq/kg, 6 Doses (Arm C): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride 55 kBq/kg IV every 28 days for up to 12 doses ("extended dose").
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
months | 13.2 [9.2 to 18.1] | 10.8 [8.1 to 13.8]
Statistical Analysis 1: Comparison: Radium-223 55 kBq/kg, 6 Doses (Arm A) vs Radium-223 88 kBq/kg, 6 Doses (Arm C); Test type: Other; p = 0.3134, Log Rank; Hazard Ratio (HR) = 1.260, 80% CI 2-sided [0.939 to 1.690] — Arm C /Arm A

5. Primary Outcome: Number of Participants With an Event Defining SSE Free Survival - Three Dose Groups As Randomized
Description: Symptomatic skeletal event (SSE) free survival is based on the following events: the use of external beam radiotherapy (EBRT) to relieve skeletal symptoms; the occurrence of new symptomatic pathological bone fractures (vertebral or nonvertebral); the occurrence of spinal cord compression; a tumor related orthopedic surgical intervention, and death.
Time Frame: as for outcome 1
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- Radium-223 55 kBq/kg, 12 Doses (Arm C): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride 55 kBq/kg IV every 28 days for up to 12 doses ("extended dose").
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
Participants | 80 | 85 | 92

6. Primary Outcome: Symptomatic Skeletal Event Free Survival - Three Dose Groups As Randomized
Description: Symptomatic skeletal event (SSE) is defined as follows: The use of external beam radiotherapy (EBRT) to relieve skeletal symptoms; The occurrence of new symptomatic pathological bone fractures (vertebral or nonvertebral); The occurrence of spinal cord compression; A tumor related orthopedic surgical intervention.
Time Frame: as for outcome 1
Population: ITT
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
months | 13.1 [11.0 to 14.6] | 12.9 [10.9 to 14.8] | 9.6 [9.0 to 10.9]

7. Secondary Outcome: Number of Participants With an Overall Survival Event - High Dose vs. Standard Dose
Description: Overall survival was defined as the time in days from the applicable start date to the date of death due to any cause. Participants who were still alive or who were lost to survival follow-up as of database cut-off date were to be censored at the last known alive date on or prior to database cut-off date.
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
Participants | 89 | 106

8. Secondary Outcome: Overall Survival - High Dose vs. Standard Dose
Description: as for outcome 7
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
months | 16.0 [14.7 to 17.2] | 14.9 [13.7 to 16.7]
Statistical Analysis 1: Comparison: Radium-223 88 kBq/kg, 6 Doses (Arm B) vs Pooled Radium-223 55 kBq/kg (Arms A and C); Test type: Other; p = 0.6205, Log Rank; Hazard Ratio (HR) = 1.075, 80% CI 2-sided [0.892 to 1.297] — Arm B/Arm (A+C)

9. Secondary Outcome: Number of Participants With an Overall Survival Event - Extended Dose vs. Standard Dose
Description: as for outcome 7
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Count of Participants; unit: Participants
Groups:
- Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A): Participants who were randomized in a 1:1:1 fashion received Xofigo (Radium-223 dichloride, BAY88-8223) 55 kBq/kg intravenously (IV) every 28 days for up to 6 doses ("standard dose").
- Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride 55 kBq/kg IV every 28 days for up to 12 doses ("extended dose").
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
Participants | 43 | 38

10. Secondary Outcome: Overall Survival - Extended Dose vs. Standard Dose
Description: as for outcome 7
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
months | 16.5 [14.0 to 19.9] | 15.2 [14.0 to 19.0]
Statistical Analysis 1: Comparison: Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) vs Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C); Test type: Other; p = 0.9958, Log Rank; Hazard Ratio (HR) = 0.999, 80% CI 2-sided [0.744 to 1.341] — Arm C/Arm A

11. Secondary Outcome: Number of Participants With an Overall Survival - Three Dose Groups As Randomized
Description: as for outcome 7
Time Frame: as for outcome 1
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
Participants | 83 | 89 | 93

12. Secondary Outcome: Overall Survival Event - Three Dose Groups as Randomized
Description: as for outcome 7
Time Frame: as for outcome 1
Population: ITT
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
months | 15.8 [14.3 to 18.1] | 16.0 [14.7 to 17.2] | 14.4 [12.1 to 16.5]

13. Secondary Outcome: Number of Participants With First Symptomatic Skeletal Event - High Dose vs. Standard Dose
Description: as for outcome 6
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
Participants | 42 | 62

14. Secondary Outcome: Time to First Symptomatic Skeletal Event - High Dose vs. Standard Dose
Description: Time to first SSE is defined as the time in days from the applicable start date to the first SSE on or following the start date.
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
months | 24.1 [18.0 to NA] — There were no sufficient events observed in this study to calculate the upper limit. | 26.3 [26.3 to NA] — There were no sufficient events observed in this study to calculate the upper limit.
Statistical Analysis 1: Comparison: Radium-223 88 kBq/kg, 6 Doses (Arm B) vs Pooled Radium-223 55 kBq/kg (Arms A and C); Test type: Other; p = 0.7461, Log Rank; Hazard Ratio (HR) = 1.068, 80% CI 2-sided [0.823 to 1.385] — Arm B/Arm (A+C)

15. Secondary Outcome: Number of Participants With First Symptomatic Skeletal Event - Extended Dose vs. Standard Dose
Description: as for outcome 6
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
Participants | 19 | 25

16. Secondary Outcome: Time to First Symptomatic Skeletal Event - Extended Dose vs. Standard Dose
Description: as for outcome 14
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
months | NA [21.2 to NA] — There were no sufficient events observed in this study to calculate the median or its upper limit of 80% CI. | 19.5 [12.3 to 23.4]
Statistical Analysis 1: Comparison: Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) vs Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C); Test type: Other; p = 0.1550, Log Rank; Hazard Ratio (HR) = 1.549, 80% CI 2-sided [1.041 to 2.306] — Arm C/Arm A

17. Secondary Outcome: Number of Participants With First Symptomatic Skeletal Event - Three Dose Groups as Randomized
Description: as for outcome 6
Time Frame: as for outcome 1
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
Participants | 37 | 42 | 48

18. Secondary Outcome: Time to First Symptomatic Skeletal Event - Three Dose Groups as Randomized
Description: as for outcome 14
Time Frame: as for outcome 1
Population: ITT
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
months | NA [26.3 to NA] — There were no sufficient events observed in this study to calculate the median or its upper limit of 80% CI. | 24.1 [18.0 to NA] — There were no sufficient events observed in this study to calculate the upper limit of 80% CI. | 18.8 [15.1 to 25.6]

19. Secondary Outcome: Number of Participants With a Radiological Progression Event-Free - High Dose vs. Standard Dose
Description: Radiological progression of soft tissue disease is determined according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 based on Magnetic resonance imaging (MRI) or computed tomography (CT) scans. Radiological progression of osseous disease is determined according to adapted PCWG2 criteria based on whole body technetium-99 bone scans. Radiological bone progression is determined if at least one of the following criteria is met: The first bone scan with ≥2 new lesions compared to baseline is observed <12 weeks from randomization and is confirmed by a second bone scan taken ≥6 weeks later showing ≥2 additional new lesions (a total of ≥4 new lesions compared to baseline); or The first bone scan with ≥2 new lesions compared to baseline is observed ≥12 weeks from randomization and the new lesions are verified on the next bone scan ≥6 weeks later (a total of ≥2 new lesions compared to baseline).
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
Participants | 77 | 141

20. Secondary Outcome: Radiological Progression Free Survival - High Dose vs. Standard Dose
Description: Radiological progression free survival is defined as the time in days from the applicable start date to the date of subsequent radiological disease progression or death from any cause (if death occurs before such progression). Participants not experiencing death or radiological disease progression as of database cut-off were censored at the last radiological disease progression assessment.
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
months | 7.5 [5.9 to 8.6] | 6.0 [5.2 to 6.2]
Statistical Analysis 1: Comparison: Radium-223 88 kBq/kg, 6 Doses (Arm B) vs Pooled Radium-223 55 kBq/kg (Arms A and C); Test type: Other; p = 0.8284, Log Rank; Hazard Ratio (HR) = 0.969, 80% CI 2-sided [0.805 to 1.167] — Arm B/Arm (A+C)

21. Secondary Outcome: Number of Participants With a Radiological Progression Event-Free - Extended Dose vs. Standard Dose
Description: Radiological progression of soft tissue disease is determined according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 based on Magnetic resonance imaging (MRI) or Computed tomography (CT) scans. Radiological progression of osseous disease is determined according to adapted PCWG2 criteria based on whole body technetium-99 bone scans.
Time Frame: as for outcome 1
Population: Baseline is randomization date
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
Participants | 49 | 47

22. Secondary Outcome: Radiological Progression Free Survival - Extended Dose vs. Standard Dose
Description: as for outcome 20
Time Frame: as for outcome 1
Population: Baseline is randomization date
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
months | 8.9 [6.3 to 11.8] | 9.0 [7.5 to 9.6]
Statistical Analysis 1: Comparison: Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) vs Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C); Test type: Other; p = 0.7896, Log Rank; Hazard Ratio (HR) = 1.059, 80% CI 2-sided [0.804 to 1.396] — Arm C/Arm A

23. Secondary Outcome: Number of Participants With a Radiological Progression Event-Free - Three Dose Groups as Randomized
Description: Radiological progression of soft tissue disease is determined according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 based on Magnetic resonance imaging (MRI) or Computed tomography (CT) scans. Radiological progression of osseous disease is determined according to adapted Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria based on whole body technetium-99 bone scans.
Time Frame: as for outcome 1
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
Participants | 77 | 77 | 90

24. Secondary Outcome: Radiological Progression Free Survival - Three Dose Groups as Randomized
Description: as for outcome 20
Time Frame: as for outcome 1
Population: ITT
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
months | 6.3 [5.1 to 7.2] | 7.5 [5.9 to 8.6] | 6.1 [5.2 to 6.6]

25. Secondary Outcome: Number of Participants With a Radiological Progression Event - High Dose vs. Standard Dose
Description: as for outcome 23
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
Participants | 63 | 115

26. Secondary Outcome: Time to Radiological Progression - High Dose vs. Standard Dose
Description: Time to radiological progression is defined as the time in days from the applicable start date to the date of subsequent radiological progression. Participants without radiological progression as of database cut-off date, whether or not surviving, were censored at the last radiological progression assessment.
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 130 | 261
months | 8.7 [6.2 to 9.7] | 6.2 [6.0 to 6.6]
Statistical Analysis 1: Comparison: Radium-223 88 kBq/kg, 6 Doses (Arm B) vs Pooled Radium-223 55 kBq/kg (Arms A and C); Test type: Other; p = 0.9274, Log Rank; Hazard Ratio (HR) = 0.986, 80% CI 2-sided [0.803 to 1.210] — Arm B/Arm (A+C)

27. Secondary Outcome: Number of Participants With a Radiological Progression Event - Extended Dose vs. Standard Dose
Description: as for outcome 20
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
Participants | 43 | 43

28. Secondary Outcome: Time to Radiological Progression - Extended Dose vs. Standard Dose
Description: as for outcome 26
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 84 | 69
months | 8.9 [6.3 to 14.6] | 9.0 [7.2 to 10.2]
Statistical Analysis 1: Comparison: Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) vs Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C); Test type: Other; p = 0.5754, Log Rank; Hazard Ratio (HR) = 1.134, 80% CI 2-sided [0.850 to 1.514] — Arm C/Arm A

29. Secondary Outcome: Number of Participants With a Radiological Progression Event - Three Dose Groups as Randomized
Description: as for outcome 20
Time Frame: as for outcome 1
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
Participants | 66 | 63 | 67

30. Secondary Outcome: Time to Radiological Progression - Three Dose Groups as Randomized
Description: as for outcome 26
Time Frame: as for outcome 1
Population: ITT
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
months | 6.2 [5.9 to 7.1] | 8.7 [6.2 to 9.7] | 6.6 [6.0 to 8.7]

31. Secondary Outcome: Timepoint Pain Improvement Rate - Three Dose Groups as Randomized
Description: Timepoint pain improvement rate is defined as the proportion of participants with a 30% and 2-point decrease in Worst pain score (WPS) from baseline over 2 consecutive assessment periods conducted at least 4 weeks apart among participants with a WPS score ≥ 4 at baseline.
Time Frame: as for outcome 1
Population: ITT
Measure: Number (80% Confidence Interval); unit: percentage
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
percentage
  Week 12 | 16.7 [10.1 to 25.7] | 16.0 [9.5 to 24.7] | 18.6 [11.1 to 28.5]
  Overall (confirmed) | 27.1 [18.7 to 37.0] | 26.0 [17.9 to 35.6] | 37.2 [27.3 to 48.1]

32. Secondary Outcome: Timepoint Pain Improvement Rate - Extended Dose vs. Standard Dose
Description: as for outcome 31
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Number (80% Confidence Interval); unit: percentage
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 22 | 20
percentage
  Week 12 | 31.8 [18.7 to 47.7] | 30.0 [16.6 to 46.7]
  Overall (confirmed) | 40.9 [26.4 to 56.8] | 55.0 [38.5 to 70.7]

33. Secondary Outcome: Number of Participants With a Pain Progression Event - High Dose vs. Standard Dose
Description: Participants were divided in 3 groups according to baseline pain evaluation: asymptomatic subjects (WPS 0 to < 1 at baseline); mildly symptomatic subjects (WPS 1-3 at baseline); and symptomatic subjects with WPS > 3 and ≤ 7 at baseline). Pain progression was defined as the occurrence of a pain increase of 2 or more points in the average (i.e., average of 7-day assessments) "worst pain in 24 hours" score from baseline observed at 2 consecutive evaluations ≥ 4 weeks apart. Participants with insufficient applicable baseline assessments or without adequate post-baseline assessments were to be censored at the applicable baseline date.
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 113 | 218
Participants | 31 | 68

34. Secondary Outcome: Time to Pain Progression - High Dose vs. Standard Dose
Description: The time to pain progression is defined for each applicable baseline for applicable participants as the time (in days) from the respective baseline until occurrence of the first post-baseline pain progression event.
Time Frame: as for outcome 1
Population: ITT. Data from Arm C are truncated at 7th dose date when pooling with Arm A.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Pooled Radium-223 55 kBq/kg (Arms A and C)
Number analyzed (Participants) | 113 | 218
months | NA [9.4 to NA] — There were no sufficient pain progression events observed in this study to calculate the median or its upper limit of 80% CI. | NA [8.6 to NA] — There were no sufficient pain progression events observed in this study to calculate the median or its upper limit of 80% CI.
Statistical Analysis 1: Comparison: Radium-223 88 kBq/kg, 6 Doses (Arm B) vs Pooled Radium-223 55 kBq/kg (Arms A and C); Test type: Other; p = 0.6214, Log Rank; Hazard Ratio (HR) = 0.898, 80% CI 2-sided [0.678 to 1.188] — Arm B/Arm (A+C)

35. Secondary Outcome: Number of Participants With a Pain Progression Event - Extended Dose vs. Standard Dose
Description: Pain progression is defined for each baseline in participants evaluable for pain progression at the applicable baseline, i.e., participants with a WPS of ≤ 7 at the respective baseline assessment.
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 78 | 65
Participants | 10 | 15

36. Secondary Outcome: Time to Pain Progression - Extended Dose vs. Standard Dose
Description: as for outcome 34
Time Frame: as for outcome 1
Population: Week 24 (W24)
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 78 | 65
months | NA [NA to NA] — There were no sufficient pain progression events observed in this study to calculate the median or its 80% CI. | NA [NA to NA] — There were no sufficient pain progression events observed in this study to calculate the median or its 80% CI.
Statistical Analysis 1: Comparison: Radium-223 Dichloride 55 kBq/kg, 6 Doses (Arm A) vs Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C); Test type: Other; p = 0.7214, Log Rank; Hazard Ratio (HR) = 0.863, 80% CI 2-sided [0.505 to 1.475] — Arm C/Arm A

37. Secondary Outcome: Number of Participants With a Pain Progression Event - Three Dose Groups as Randomized
Description: as for outcome 35
Time Frame: as for outcome 1
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 110 | 113 | 108
Participants | 32 | 31 | 46

38. Secondary Outcome: Time to Pain Progression - Three Dose Groups as Randomized
Description: as for outcome 34
Time Frame: as for outcome 1
Population: ITT
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 110 | 113 | 108
months | NA [8.9 to NA] — There were no sufficient pain progression events observed in this study to calculate the median or its upper limit of 80% CI. | NA [9.4 to NA] — There were no sufficient pain progression events observed in this study to calculate the median or its upper limit of 80% CI. | 10.1 [8.8 to 11.8]

39. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events are events starting or worsening from the initiation of treatment until 30 days after the last administration of radium-223 dichloride. The intensity of an AE is classified according to the grades specified by the National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE).
Time Frame: as for outcome 1
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 124 | 121 | 125
Participants
  Any TEAE | 118 | 119 | 116
  Grade 1 | 23 | 20 | 18
  Grade 2 | 52 | 40 | 34
  Grade 3 | 38 | 46 | 49
  Grade 4 | 4 | 11 | 11
  Grade 5 | 1 | 2 | 4
  Serious | 25 | 36 | 37
  Any drug-related TEAE | 73 | 73 | 57

40. Other Pre Specified Outcome: Number of Participants With Change in Analgesic Use From Baseline to Worst Status Post-Baseline
Description: Analgesic use in this study were captured via two methods: Analgesic concomitant medication case report form, where the physician records the analgesic medication prescribed to manage pain; 24 hour analgesic consumption case report form, in which all analgesic medication taken in the last 24 hours.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223 55 kBq/kg, 6 Doses (Arm A) | Radium-223 88 kBq/kg, 6 Doses (Arm B) | Radium-223 Dichloride 55 kBq/kg, 12 Doses (Arm C)
Number analyzed (Participants) | 130 | 130 | 131
Participants
  Strong Opioid - No Change | 22 | 27 | 26
  From Strong Opioid to Weak Opioid | 1 | 0 | 2
  From Strong Opioid to No analgesic or Non-opioid | 18 | 9 | 13
  From Strong Opioid to Missing | 2 | 0 | 4
  From No analgesic or Non-opioid to Strong Opioid | 24 | 26 | 25
  From No analgesic or Non-opioid to Weak Opioid | 5 | 8 | 12
  No analgesic or Non-opioid - No Change | 46 | 41 | 30
  From No analgesic or Non-opioid to Missing | 5 | 5 | 5

ADVERSE EVENTS:
Time Frame: From starting of study medication over a period of approximately 3 years since first participant was enrolled.
Groups:
- Radium-223 55 kBq/kg Arm A (6 Doses): Participants who were randomized in a 1:1:1 fashion received Xofigo (Radium-223 dichloride, BAY88-8223) 55 kBq/kg intravenously (IV) every 28 days for up to 6 doses ("standard dose").
- Radium-223 88 kBq/kg Arm B (6 Doses): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride (Xofigo, BAY88-8223) 88 kBq/kg IV every 28 days for up to 6 doses ("high dose").
- Radium-223 55 kBq/kg Arm C (12 Doses): Participants who were randomized in a 1:1:1 fashion received Radium-223 dichloride (Xofigo, BAY88-8223) 55 kBq/kg IV every 28 days for up to 12 doses ("extended dose").
Arm/Group | Radium-223 55 kBq/kg Arm A (6 Doses) | Radium-223 88 kBq/kg Arm B (6 Doses) | Radium-223 55 kBq/kg Arm C (12 Doses)
All-Cause Mortality (participants affected / at risk) | 98/125 | 100/124 | 102/121
Serious Adverse Events (participants affected / at risk) | 25/125 | 36/124 | 37/121
Other Adverse Events (participants affected / at risk) | 109/125 | 111/124 | 111/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 55 kBq/kg Arm A (6 Doses) (N=125) | Radium-223 88 kBq/kg Arm B (6 Doses) (N=124) | Radium-223 55 kBq/kg Arm C (12 Doses) (N=121)
Anaemia (Blood and lymphatic system disorders) | 3 (7) | 6 (24) | 4 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (13) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (28) | 2 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 2 (3) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (2) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 1 (1)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 1 (2)
Alcohol intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (10) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (4)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 6 (7) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radium-223 55 kBq/kg Arm A (6 Doses) (N=125) | Radium-223 88 kBq/kg Arm B (6 Doses) (N=124) | Radium-223 55 kBq/kg Arm C (12 Doses) (N=121)
Anaemia (Blood and lymphatic system disorders) | 29 (64) | 33 (69) | 30 (79)
Neutropenia (Blood and lymphatic system disorders) | 2 (7) | 10 (21) | 5 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (14) | 10 (26) | 10 (33)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3) | 10 (12)
Constipation (Gastrointestinal disorders) | 21 (27) | 10 (11) | 18 (20)
Diarrhoea (Gastrointestinal disorders) | 26 (34) | 28 (39) | 26 (32)
Nausea (Gastrointestinal disorders) | 31 (38) | 29 (33) | 28 (39)
Vomiting (Gastrointestinal disorders) | 12 (16) | 15 (19) | 17 (22)
Asthenia (General disorders) | 12 (15) | 9 (11) | 17 (25)
Fatigue (General disorders) | 39 (58) | 37 (46) | 35 (49)
Oedema peripheral (General disorders) | 9 (10) | 6 (6) | 7 (7)
Pyrexia (General disorders) | 4 (4) | 9 (9) | 5 (5)
Urinary tract infection (Infections and infestations) | 2 (2) | 7 (7) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 9 (14) | 4 (4)
Neutrophil count decreased (Investigations) | 4 (6) | 9 (22) | 3 (11)
Weight decreased (Investigations) | 12 (17) | 6 (7) | 19 (24)
Decreased appetite (Metabolism and nutrition disorders) | 31 (39) | 24 (25) | 26 (31)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (26) | 17 (22) | 19 (24)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (25) | 18 (19) | 24 (29)
Bone pain (Musculoskeletal and connective tissue disorders) | 23 (26) | 19 (21) | 27 (32)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (8) | 8 (8) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 7 (7) | 11 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (9) | 4 (4) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (15) | 9 (10) | 12 (13)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 7 (9)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 (15) | 5 (7) | 8 (9)
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 1 (1) | 7 (12)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3) | 8 (10)
Headache (Nervous system disorders) | 7 (8) | 6 (7) | 6 (7)
Depression (Psychiatric disorders) | 4 (5) | 1 (1) | 7 (7)
Insomnia (Psychiatric disorders) | 9 (9) | 6 (7) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 4 (4) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 7 (7)
Hypertension (Vascular disorders) | 6 (7) | 5 (9) | 7 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12-18 months after database lock at the earliest. Bayer will have 30-45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable). No publication of single center data should be done prior of publication if multi-center data.

DOCUMENTS (2):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT02023697/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT02023697/SAP_003.pdf